CLINICAL TRIAL: NCT02627352
Title: Prospective Evaluation of the New Micropulse Transscleral Cyclophotocoagulation
Brief Title: How Safe and Effective is Micropulse Transscleral Cyclophotocoagulation in Patients With Uncontrolled Glaucoma?
Acronym: TSCPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Marlene Moster, MD, Principal Investigator, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-439
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; Micropulse Transscleral Cyclophotocoagulation; Intraocular Pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Diode Laser Cyclophotocoagulation
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transscleral Cyclophotocoagulation (Experimental): Subjects undergo a Micropulse Transscleral Cyclophotocoagulation(TSCPC) laser surgery, where a diode laser is used to damage tissue of the ciliary body, the tissue inside the eye that produces aqueous, the clear fluid in the eye that maintains intraocular pressure. This causes it to produce less aqueous.
  Interventions: Procedure: Micropulse Transscleral Cyclophotocoagulation

INTERVENTIONS:
Procedure: Micropulse Transscleral Cyclophotocoagulation — In mTSCPC, a diode laser is used to damage tissue of the ciliary body, the tissue inside the eye that produces aqueous, the clear fluid in the eye that maintains intraocular pressure. This causes it to produce less aqueous.
  Other Names: mTSCPC

SUMMARY:
The purpose of this study is to investigate the surgical outcomes of the micropulse transscleral cyclophotocoagulation (mTSCPC) in patients with uncontrolled glaucoma; analyze intraocular pressure lowering effect; and correlate related treatment parameters pending enrollment of sufficient numbers of dark pigmented versus light pigmented eyes.

DETAILED DESCRIPTION:
If the subject agrees to participate in this study, he/she will come in for a screening visit to make sure they qualify for the study. Following the surgical procedure, principal investigator will perform a standard postoperative examination at Day 1, Week 1, Month

1, Month 3, Month 6 and Month 12, in addition to any other visits the investigator feels may be necessary.

Screening Visit: At the screening visit, the subjects medical history and current medications will be reviewed. Pre-operative eye pressure and visual acuity will be noted. The Kowa Flare Meter-500 laser flare meter and slit lamp (the table-top microscope used for examining the eye) will be used to measure inflammation in subjects anterior chamber (the fluid-filled space between the iris (colored part of the eye) and cornea (clear front part of the eye that covers the iris and pupil).

Surgery: On the day of the subjects surgery, the subject will undergo the standard procedure for transscleral cyclophotocoagulation (TSCPC) laser surgery using the micropulse delivery mode of diode laser. After the Principal investigator finishes with the laser, he/she will perform anterior chamber paracentesis, which will help reduce the pressure in the subjects eye quickly and temporarily. To do this, the principal investigator will puncture the cornea (the clear front part of the eye that transmits and focuses light into the eye) to remove some of the aqueous (fluid inside the eye). Paracentesis is usually not done if TSCPC is performed using the "continuous" delivery mode.

Post-Operative Exams: At each of the post-operative office visits (Day 1, Week 1, Months 1, 3, 6 and 12) a detailed medical/eye history will be taken, including all current medications, vision will be tested and an eye examination will be performed, including measurement of eye pressure. Subject will be asked about his/her comfort level in regards to pain. At visit Day 1 and Month 1 the amount of anterior chamber inflammation will again be measured (as described in Screening Visit).

ELIGIBILITY:
Inclusion Criteria: Patients with a minimum of 6 months follow-up with uncontrolled glaucoma as defined by:

* Progression and/or intraocular pressure above target despite maximal tolerated medical therapy
* Evidence of glaucomatous optic nerve damage and glaucomatous visual field loss in at least one hemifield

Exclusion Criteria:

* Age ≤ 20 years old.
* Patients who had undergone previous intraocular surgery or ocular laser treatment within 2 months of enrolment.
* Patients who had undergone previous conventional continuous wave mode TSCPC within 1 months of enrolment.
* Patients with significant scleral thinning as defined by greater than 1 clock hour.
* Patients with any medical condition that would preclude the subject from providing informed consent or reliable and valid data.
* Patients enrolled in other prospective clinical trials.
* Albino patients that have no pigmentation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure-lowering effect | 2 years
  The primary outcome measure will be treatment success, defined by an intraocular pressure (IOP) between 5 and 21mmHg (millimeters of mercury) or a 20% reduction from baseline with or without the addition of anti-glaucoma medications. Within the success group there will be sub-categories of ''qualified success" defined as achieving target IOP with the aid of anti-glaucoma medications.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene R Moster, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Institute, Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript has been submitted for publication.